CLINICAL TRIAL: NCT04519008
Title: Effectiveness and Security Testing of a Mobile App (B·RIGHT) for Adolescents With Attention-Deficit/Hyperactivity Disorder and Emotion Dysregulation
Brief Title: Effectiveness and Security Testing of a Mobile App
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 51/20
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual plus mobile app (Experimental): Those who will receive naturalistic treatment in outpatient setting and also the mobile app
  Interventions: Device: Mobile app; Combination Product: Treatment as usual
- Treatment as usual (Active Comparator): Those who will receive naturalistic treatment in outpatient setting but not the mobile app
  Interventions: Combination Product: Treatment as usual

INTERVENTIONS:
Device: Mobile app — Medical device for improving emotion dysregulation
  Arms: Treatment as usual plus mobile app
Combination Product: Treatment as usual — Bimonthly individual psychotherapy and psychostimulant medications

SUMMARY:
To assess the effectiveness and security of a mobile App (beta version) for self-managing emotion dysregulation in a pragmatic randomized controlled trial with 80 adolescents with attention-deficit/hyperactivity disorder comparing 40 patients with treatment as usual (TAU) with 40 patients with TAU plus the mobile App

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) of attention-deficit/hyperactivity disorder
* High emotion dysregulation severity
* Aged 14 to 17 years
* Outpatient setting (Consorci Sanitari del Maresme

Exclusion Criteria:

* Comorbidity with mental retardation
* Comorbidity with psychotic disorder
* Comorbidity with autism spectrum disorder

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Emotion dysregulation severity | 9 months
  Severity of emotional dysregulation as measured by a single score from the The DERS (Difficulties in Emotion Regulation Scale) (range: 0-88; the higher the score, the more severe the emotion dysregulation severity).
Smartphone addiction | 9.months
  Severity of smartphone addiction as measured by the Spanish version of the The Smartphone Addiction Scale (SAS) (range: 10-60; the higher the score, the more severe the smartphone addiction severity).